CLINICAL TRIAL: NCT03962998
Title: A Randomized Unblinded Feasibility Study Evaluating the Use of Oral Administration of MB-102 Versus Dual Sugar Testing for Gut Permeability in Normal Subjects and Subjects With Active Small Bowel Crohn's Disease
Brief Title: Oral Administration of MB-102 Versus Dual Sugar Testing for Gut Permeability
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: MediBeacon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MB-300-01
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Crohn Disease
Keywords: Gut permeability; Intestinal permeability; MB-102
MeSH Terms: conditions — Crohn Disease | interventions — Lactulose; relmapirazin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lactulose/Rhamnose (Active Comparator): 1000 mg of lactulose and 200 mg of rhamnose administered orally as a 10 mL solution
  Interventions: Drug: Lactulose/Rhamnose solution
- MB-102 (Experimental): 4 μmol of MB-102/kg body weight administered orally as a solution
  Interventions: Drug: MB-102

INTERVENTIONS:
Drug: Lactulose/Rhamnose solution — Lactulose/Rhamnose solution administered orally followed by measurement of excreted lactulose and rhamnose in urine
  Arms: Lactulose/Rhamnose
Drug: MB-102 — MB-102 solution administered orally followed by measurement of excreted MB-102 in urine
  Arms: MB-102

SUMMARY:
The objectives of the study are to evaluate the safety and tolerability of oral administration of MB-102, and to evaluate the use of MB-102 as a means of measuring gut permeability in normal participants (n=10) and in those with radiologic evidence of small bowel Crohn's disease (n=10).

DETAILED DESCRIPTION:
This study is a single center, randomized, open label, cross-over study evaluating MB-102 versus dual sugar testing using lactulose and rhamnose for the assessment of gut permeability. Participants will be screened within 30 days of Day 1, and eligible participants will be randomized to receive either an oral dose of MB-102 or the dual sugar test on Day 1. At a second study visit occurring between 3 to 7 days after completion of the first test, participants will return to the study center for the second test. Following completion of the second test, participants will return to the study center 7 ±3 days for a follow-up visit to evaluate safety.

ELIGIBILITY:
Inclusion criteria for all participants:

* Age > 18 years - male or non-pregnant or lactating females
* Participants willing to comply with study requirements
* Participants who have signed an informed consent form
* Normal or non-clinically significant screening and baseline 12 lead electrocardiogram (ECG) in the opinion of the principal investigator (PI)
* Estimated glomerulofiltration rate (eGFR) > 75 mL/min/1.73 m^2
* Agreement to not utilize nonsteroidal anti-inflammatory drugs (NSAIDs) until study completion.

Inclusion criteria for participants with Crohn's disease:

* Participants with active small bowel Crohn's disease diagnosed by an abnormal Magnetic Resonance Enterography (MRE) within 1 month prior to screening
* Active Crohn's disease must be characterized by mucosal hyperemia, and/or bowel wall thickening and/or vascular engorgement

Exclusion criteria for all participants:

* Women who are pregnant, lactating, or planning to become pregnant during the study, or women who are of childbearing potential unwilling to use an adequate method of birth control a. Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 7 days post dose
* Participation in another interventional trial within 30 days of dosing or concurrently enrolled in any other medical research study which could impact the results of the study
* Unable to tolerate an overnight fast
* NSAID use within 14 days of Day 1
* History of drug or alcohol abuse within the past year
* Diagnosis of ulcerative colitis, indeterminate colitis, pseudomembranous colitis, or celiac disease
* Prior or current diagnosis of an autoimmune disease
* Gastrointestinal surgery (including appendectomy) within 12 weeks prior to screening or has surgery planned or deemed likely to require surgery during the study
* Type 1 or 2 diabetes
* History of severe allergic hypersensitivity reactions (unacceptable adverse events) or anaphylactoid reaction to any allergen including drugs, or MB-102 (intolerance to a drug is not considered a drug allergy)
* Known history of testing positive for acquired immunodeficiency syndrome (AIDS) or human immunodeficiency virus (HIV)
* Site personnel immediately associated with the study or their immediate family members
* Any characteristics which, in the opinion of the investigator, makes the participant a poor candidate for participation in the clinical trial
* Prior exposure to MB-102
* Any changes to chronic medication therapy or initiation of new medications between Testing Day 1 and Testing Day 2
* Current urinary tract infection
* Body mass index > 30 kg/m^2
* Prior history of small bowel malignancy or resection surgery
* Unable to meet the requirements of the study including 12+ hour study visits

Additional exclusion criteria for normal participants:

* Fecal transplant within 1 year
* Prior or current graft-vs.-host disease
* Prior or current history of diverticulitis
* Current or prior history of fatty liver
* Current use of any biologic therapy or current use of the following medications: sulfasalazine, mesalamine, olsalazine, balsalazide, prednisone, cyclosporine, azathioprine, 6-mercaptopurine, tacrolimus, methotrexate, intravenous immunoglobulin, anti-diarrheal agents
* Prior antibiotic therapy within 30 days of screening
* Undiagnosed chronic gastrointestinal upset or food intolerance history
* Recent history of significant unplanned weight loss, blood in the stool or acute episodes of diarrhea
* First-degree relative (sibling, parent, child) has inflammatory bowel disease (Crohn's disease, ulcerative colitis, proctitis, indeterminate colitis)
* History of Crohn's disease

Additional exclusion criterion for participants with Crohn's disease:

- Participant on Total Parenteral Nutrition (TPN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Mean urine concentration of MB-102 over time in normal participants and in those with Crohn's disease | Pre-dose and 1, 2, 4, 6, 8, 10, and 12 hours
  Urine samples will be collected pre-dose (time 0), each time the participant voids, and at the protocol-defined time points after oral administration of MB-102. The total volume of urine excreted will be recorded. Urine samples will be analyzed using validated analytical methods.

SECONDARY OUTCOMES:
Correlation between MB-102 excretion and the results of dual sugar testing in normal participants and in those with Crohn's disease | Pre-dose and 1, 2, 4, 6, 8, 10, and 12 hours
  For MB-102 excretion evaluation, urine samples will be collected pre-dose (time 0), each time the participant voids, and at the protocol-defined time points after oral administration of MB-102. The total volume of urine excreted will be recorded. Urine samples will be analyzed using validated analytical methods. For the dual sugar test, participants will consume a 10 mL solution (1000 mg of lactulose and 200 mg of rhamnose). Urine will be collected pre-dose (time 0), each time the participant voids, and at the protocol-defined time points after consuming the sugar solution. The total volume of urine excreted will be recorded. Urine samples will be analyzed using validated analytical methods.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Dorshow, PhD, Study Director — MediBeacon
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No